CLINICAL TRIAL: NCT02720211
Title: Spectacle Tints and Thin-Films to Reduce Headache Frequency in Patients With Chronic Migraine
Brief Title: Spectacle Tints and Thin-Films for Migraine
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Too difficult to enroll according to inclusion/exclusion criteria
Sponsor: University of Utah (Other)
Collaborators: Axon Optics, LLC (Industry); Mayo Clinic (Other); Brigham and Women's Hospital (Other); Northwell Health (Other)
Responsible Party: Principal Investigator, Bradley Katz, MD, PhD, University of Utah
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB #86498
Record Dates: First submitted 2016-03-21; First posted 2016-03-25 (Estimated); Results first posted 2022-11-29 (Actual); Last update posted 2022-11-29 (Actual); Status verified 2022-11

CONDITIONS: Headache Migraine Chronic
Keywords: headache; photophobia; migraine; light sensitivity; tints; thin films
MeSH Terms: conditions — Headache; Photophobia; Migraine Disorders

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Gray tinted spectacle lenses (Active Comparator): Subjects in this arm will be asked to wear a neutral gray tint that blocks all wavelengths equally
  Interventions: Device: Gray tinted spectacle lenses
- Thin-Film spectacle lenses (Experimental): Subjects in this arm well be asked to wear a thin-film coating that specifically blocks 480-nm wavelength
  Interventions: Device: Thin-Film spectacle lenses

INTERVENTIONS:
Device: Gray tinted spectacle lenses — A neutral gray optical tint designed to block all wavelengths in the visible spectrum
  Arms: Gray tinted spectacle lenses
Device: Thin-Film spectacle lenses — A thin film optical notch filter designed to block 480-nm light in the visible spectrum
  Arms: Thin-Film spectacle lenses

SUMMARY:
Nearly all migraine sufferers report sensitivity to light during a headache and a significant proportion of sufferers report light sensitivity between attacks. Light is also a common trigger for migraine headaches. Spectacle lenses that have been treated with tints and spectacle lenses that have been treated with thin-films have both been shown to reduce light sensitivity and headache in patients with migraine. At this time, it is not clear which spectacle lens treatment is superior. The purpose of this trial is to determine if there's a significant, therapeutic advantage to either spectacle lens treatment. Both treatments could be a novel, non-invasive adjuvant in the treatment of migraine.

DETAILED DESCRIPTION:
Approximately 6% of men and 18% of women are afflicted with migraines. (Stovner et al., 2006) Over 90% of patients with migraines report a sensitivity to light (photophobia) during headaches. (Evans et al., 2008) Some migraine sufferers report that light can trigger a migraine and some have a chronic sensitivity to light (Main et al., 1997). Migraineurs are especially sensitive to non-incandescent lighting sources such as fluorescent lights, computer monitors, and gas-vapor lamps (Katz and Digre, 2016).

The pathway that mediates photophobia appears to involve intrinsically photosensitive retinal ganglion cells ("IPRGCs"; Hattar et al., 2002) and trigeminal afferents (Noseda et al., 2010; Digre and Brennan, 2012). These retinal cells do not require input from photoreceptors to be activated by light, and they have been shown to be responsible for circadian rhythm entrainment and the pupillary light reflex. As such, these cells constitute a pathway separate from that of the visual pathway (Güler et al., 2008). IPRGCs contain the chromophore melanopsin. In these cells, 480 nm light (in the blue-green portion of the visible spectrum) isomerizes melanopsin and triggers the phototransduction cascade. However, IPRGCs can also be stimulated by rods and cones. Thus, IPRGCs can be stimulated directly by 480-nm light or indirectly by any light in the visible spectrum.

In the present study, the investigators will use a neutral gray tint to decrease stimulation of the eye by all wavelengths in the visible spectrum. The investigators will compare this intervention to a thin-film spectacle coating designed to specifically block 480-nm light. The gray tint will decrease both direct and indirect stimulation of the IPRGCs by blocking all wavelengths of the visible spectrum. The 480-nm thin-film will specifically target direct stimulation of the IPRGC.

All tints and thin films will be calibrated such that the optical density, that is the overall "darkness" of all study lenses, will be the same. All study lenses will appear to have the same overall light blocking effect to study subjects. The lenses are intended to be a preventative or prophylactic treatment for chronic migraine.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet the International Headache Society criteria for chronic migraine (International Classification of Headache Disorders, 3rd edition (Headache Classification Committee of the International Headache Society, 2013). All subjects must be between the ages of 18 and 60 years-old.

To be included in the study, in the best judgment of the investigator, subjects must be stable on their current migraine treatment regimen. Stability is defined as no major changes in therapy contemplated within the next 4 months.

Exclusion Criteria:

* Subjects with other light sensitive conditions, such as iritis and blepharospasm, will be excluded. Subjects with best-corrected visual acuity less than 20/40 will be excluded. Subjects with diseases of the retina, such as diabetic retinopathy and macular degeneration will be excluded. Subjects using medications known to affect the eye will be excluded (e.g. chloroquine, hydroxychloroquine, ethambutol, amiodarone). Due to constraints on the manufacture and mounting of study lenses into study frames, the study must exclude subjects who are very nearsighted (more than 4 diopters), subjects who are very farsighted (more than 2 diopters), and subjects who have more than 2.5 diopters of astigmatism.

Because of the cyclical effects of botulinum toxin injections and other nerve blocks, patients undergoing these treatments will be excluded. Subjects must not have had any injections or blocks within 4 months of enrollment and should not receive any further blocks until they exit the study.

Subjects with continuous daily headache (a headache frequency of 100%) will be excluded. Subjects who do not have a headache frequency of at least 50% will be excluded.

Subjects with medication overuse headache will be excluded. A patient with a history of medication overuse who has not overused abortive medications for the past 4 months can be included.

Subjects who abuse alcohol or use illicit drugs will be excluded. Subjects considered to be from vulnerable populations will be excluded, including pregnant women, prisoners, subject who are mentally disabled, subjects with cognitive or decisional impairment, and wards of the state

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-11-06 (Actual); Study Completion 2018-11-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bradley Katz, MD, Principal Investigator — Axon Optics, LLC
Locations (4):
- United States (4):
  - Mayo Clinic, Phoenix, Arizona
  - Brigham and Women's Hospital; John R Graham Headache Center; Harvard University,, Boston, Massachusetts
  - Headache Center of the Neuroscience Institute; Hofstra Northwell Health; Northshore University Hospital, Great Neck, New York
  - John A Moran Eye Center; University of Utah Hospitals and Clinics, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Gray Tinted Spectacle Lenses | Thin-Film Spectacle Lenses
Started | 5 | 5
Completed | 5 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Gray Tinted Spectacle Lenses: Subjects in this arm will be asked to wear a neutral gray tint that blocks all wavelengths equally
  Thin-Film spectacle lenses: A thin film optical notch filter designed to block 480-nm light in the visible spectrum
- Thin-Film Spectacle Lenses: Subjects in this arm well be asked to wear a thin-film coating that specifically blocks 480-nm wavelength
  Gray tinted spectacle lenses: A neutral gray optical tint designed to block all wavelengths in the visible spectrum
- Total: Total of all reporting groups
Arm/Group | Gray Tinted Spectacle Lenses | Thin-Film Spectacle Lenses | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Continuous [Mean (Full Range); unit: years] | 40 [20 to 60] | 40 [20 to 60] | 40 [20 to 60]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 4 | 8
  Male | 1 | 1 | 2
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Headache Frequency
Description: average number of days (in one month) with at least one headache lasting at least 4 hours
Time Frame: one month
Measure: Mean (Standard Error); unit: days
Arm/Group | Gray Tinted Spectacle Lenses | Thin-Film Spectacle Lenses
Number analyzed (Participants) | 5 | 5
days | 12 (1.0) | 15 (1.5)

2. Secondary Outcome: Headache Impact
Description: Headache impact as measured by the headache impact test (HIT-6) HIT-6 total score range between 36 and 78, with larger scores reflecting greater impact Scores less than or equal to 49 = Little or no impact Scores between 50 and 55 = Some impact Scores between 56 and 59 = Substantial impact Scores 60 or great = Severe impact
Time Frame: one month
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Gray Tinted Spectacle Lenses | Thin-Film Spectacle Lenses
Number analyzed (Participants) | 5 | 5
score on a scale | 50 (5) | 55 (5)

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: no difference
Arm/Group | Gray Tinted Spectacle Lenses | Thin-Film Spectacle Lenses
All-Cause Mortality (participants affected / at risk) | 0/5 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2018-04-18): https://cdn.clinicaltrials.gov/large-docs/11/NCT02720211/Prot_SAP_000.pdf
  • Informed Consent Form (2018-04-18): https://cdn.clinicaltrials.gov/large-docs/11/NCT02720211/ICF_001.pdf